CLINICAL TRIAL: NCT01454089
Title: A Randomized, Double-blind Phase 2 Study Comparing Gemcitabine and Cisplatin in Combination With OGX-427 or Placebo in Patients With Advanced Transitional Cell Carcinoma
Brief Title: A Phase 2 Study Comparing Chemotherapy in Combination With OGX-427 or Placebo in Patients With Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OGX-427-02
Record Dates: First submitted 2011-10-05; First posted 2011-10-18 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Urologic Neoplasms; Metastatic Bladder Cancer; Urinary Tract Neoplasms
Keywords: bladder; urinary tract; transitional cell carcinoma; metastatic bladder cancer; chemotherapy
MeSH Terms: conditions — Urologic Neoplasms; Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — apatorsen; Gemcitabine; Cisplatin; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- OGX-427 600 mg (Experimental): Standard chemotherapy (gemcitabine and cisplatin) in combination with OGX-427 (600 mg)
  Interventions: Drug: OGX-427 600 mg; Drug: Gemcitabine; Drug: Cisplatin; Drug: Carboplatin
- OGX-427 1000 mg (Experimental): Standard chemotherapy (gemcitabine and cisplatin) in combination with OGX-427 (1000 mg)
  Interventions: Drug: OGX-427 1000 mg; Drug: Gemcitabine; Drug: Cisplatin; Drug: Carboplatin
- Placebo (Active Comparator): Standard chemotherapy (gemcitabine and cisplatin) in combination with placebo
  Interventions: Drug: Placebo; Drug: Gemcitabine; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: OGX-427 600 mg — Patients will receive three loading doses of 600 mg Study Drug within a 9-day period. Following the loading dose period, patients will receive weekly Study Drug infusions (600 mg IV) on Days 1, 8 and 15 of each 21-day cycle.
  Other Names: apatorsen
  Arms: OGX-427 600 mg
Drug: OGX-427 1000 mg — Patients will receive three loading doses of 600 mg Study Drug within a 9-day period. Following the loading dose period, patients will receive weekly Study Drug infusions (1000 mg IV) on Days 1, 8 and 15 of each 21-day cycle.
  Other Names: apatorsen
  Arms: OGX-427 1000 mg
Drug: Placebo — Patients will receive three loading doses of placebo within a 9-day period. Following the loading dose period, patients will receive weekly placebo infusions (IV) on Days 1, 8 and 15 of each 21-day cycle.
  Arms: Placebo
Drug: Gemcitabine — Patients will receive gemcitabine (1000 mg/m^2) for up to 6 cycles administered IV on Days 1 and 8 of each 21-day cycle following Study Drug infusion. The Cycle 1, Day 1 administration of chemotherapy must occur within 5 days of the third loading dose of Study Drug.
Drug: Cisplatin — Following the administration of gemcitabine on Day 1, cisplatin (70 mg/m^2) will be administered IV for up to 6 cycles. The Cycle 1, Day 1 administration of chemotherapy must occur within 5 days of the third loading dose of Study Drug.
Drug: Carboplatin — Following the administration of gemcitabine on Day 1, cisplatin (70 mg/m^2) is to be administered IV for up to 6 cycles; however, carboplatin could be substituted for cisplatin for some unacceptable toxicities. The Cycle 1, Day 1 administration of chemotherapy must occur within 5 days of the third loading dose of Study Drug.

SUMMARY:
The primary objective of this study is to ascertain whether there is evidence of longer survival relative to the control arm for three comparisons: 600 mg OGX-427 Arm to control Arm; 1000 mg OGX-427 Arm to control Arm; and pooled 600 mg and 1000 mg OGX-427 Arms to control Arm.

DETAILED DESCRIPTION:
Following 3 loading doses, participants receive chemotherapy and study drug on a 21-day cycle during the Treatment Period (Chemotherapy Period) until disease progression, completion of 6 cycles, toxicity or voluntary participant withdrawal. Participants who do not have documented disease progression and have completed a minimum of four cycles of chemotherapy continue to receive weekly Study Drug maintenance therapy during the Maintenance Period until disease progression or the participant fulfills one of the other reasons for withdrawal from protocol treatment, unless they have been discontinued from protocol treatment for unacceptable toxicity related to study drug. All participants have an End of Treatment (EOT) visit when they are withdrawn from all study treatment (chemotherapy and maintenance). All participants are followed until documented disease progression. Once disease progression is documented, participants enter a Survival Follow-up Period during which data are collected regarding further cancer therapy, secondary malignancy, and survival status.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of consent
2. Histologically documented metastatic or locally inoperable advanced transitional cell carcinoma (TCC) of the urinary tract (bladder, urethra, ureter and renal pelvis) (T4b, N2, N3 or M1 disease) NOTE: Certain mixed histologies that are predominately (≥ 50%) TCC are eligible: squamous, adenocarcinoma, and undifferentiated. Mixed undifferentiated histology requires immunohistochemistry (IHC) consistent with a TCC origin. Mixed small-cell histologies are excluded
3. Measurable disease defined as at least one target lesion that has not been irradiated and can be accurately measured in at least one dimension by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
4. No prior systemic chemotherapy with the following exceptions:

   * Prior use of radiosensitizing single agent therapy is allowed
   * Prior neoadjuvant and adjuvant chemotherapy may be allowed
5. Minimum of 21 days since prior major surgery or radiation therapy
6. Karnofsky performance status ≥ 70%
7. Required laboratory values at baseline:

   * absolute neutrophil count (ANC) ≥ 1.5 x 10^9 cells/L
   * platelet count ≥ 125 x 10^9/L
   * calculated creatinine clearance ≥ 60 mL/minute
   * bilirubin ≤ 1.5 x upper limit of normal (ULN; ≤ 2.5 x ULN if secondary to Gilbert's disease)
   * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x ULN
8. If of child-bearing potential, willing to use contraceptives
9. Willing to give written informed consent

Exclusion Criteria:

1. A candidate for potential curative surgery or radiotherapy
2. Intravesical therapy within the last 3 months
3. Documented brain metastasis or carcinomatous meningitis, treated or untreated. NOTE: Brain imaging is not required unless the patient has symptoms or physical signs of central nervous system (CNS) disease.
4. Peripheral neuropathy ≥ Grade 2
5. Known serious hypersensitivity to gemcitabine, cisplatin or carboplatin
6. Current serious, uncontrolled medical condition such as congestive heart failure, angina, hypertension, arrhythmia, diabetes mellitus, infection, etc. or any condition such as a psychiatric illness which in the opinion of the investigator would make the patient unacceptable for the protocol
7. Cerebrovascular accident, myocardial infarction or pulmonary embolus within 6 months of randomization
8. Active second malignancy (except non-melanomatous skin cancer): active secondary malignancy is defined as a current need for cancer therapy or a high possibility (> 30%) of recurrence during the study
9. Pregnant or nursing (must have a negative serum or urine pregnancy test within 72 hours prior to randomization)
10. Participating in a concurrent clinical trial of an experimental drug, vaccine or device. Participation in an observational study is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2011-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Baseline to date of death by any cause (up to approximately 12 months)
  OS is defined as the time from randomization to death from any cause; OS was censored on date of last contact for participants still alive at time of analysis.

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (AEs), Serious AEs, and Grade 3 or Higher AEs | From initiation of study drug to end of study (up to 8 months)
  Treatment-emergent AEs are defined as and AE that occurred after the first dose of study drug up to 30 days after the last dose of study drug. AEs were graded using National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Treatment-emergent AEs could have occurred during loading dose period, chemotherapy period, maintenance period, and treatment period A detailed summary of adverse events is located in the Reported Adverse Event Module.
Number of Participants With ≥ 1 Hematology Abnormality and ≥ 1 Grade 3 or Higher Hematology Abnormality | Screening through End of Study Visit (Within 30 [±7] days following withdrawal of study treatment)
Number of Participants With ≥ 1 Chemistry Laboratory Abnormality and ≥ 1 Grade 3 or Higher Chemistry Laboratory Abnormality | Screening through End of Study Visit (Within 30 [±7] days following withdrawal of study treatment)
Number of Participants With ≥ 1 Urinalysis Abnormality and ≥ 1 Grade 3 or Higher Urinalysis Abnormality | Screening through End of Study Visit (Within 30 [±7] days following withdrawal of study treatment)
Best Objective Tumor Response | Baseline to measured progressive disease (up to approximately 12 months)
  Complete Response (CR): Complete disappearance of all measurable and non-measurable disease with no new lesions. Any pathological lymph node (target or non-target) must have a reduction in short axis to < 10 mm). All markers of disease must have normalized. Partial Response (PR): A decrease from baseline of ≥ 30% of the diameter(s) of all target measurable lesions with no unequivocal progression of non-measurable lesions and no new lesions. Stable Disease (SD): Does not qualify for CR, PR, or progression. Disease Progression (PD): If at least one of following criteria is met: 1. Appearance of any new lesion or site of disease. 2. A 20% increase in the sum of the diameter(s) of target measurable lesions over either the smallest sum observed or over baseline if no decrease during therapy has occurred. The sum must also demonstrate an absolute increase of at least 5 mm. 3. Unequivocal progression of non-target lesions alone.
Overall Response Rate (ORR) and Disease Control Rate | Baseline to measured progressive disease (up to approximately 12 months)
  Participants were defined as having an "overall response" if their best response is either confirmed CR, confirmed PR, unconfirmed CR or unconfirmed PR. ORR was defined as the percent of participants who had an overall response. Participants were defined as having "disease control" if their best response is confirmed CR, confirmed PR, unconfirmed CR, unconfirmed PR or SD. The disease control rate (DCR) was defined as the percent of participants with disease control. (See "Best Objective Tumor Response" Outcome Measure above for response category definitions.)
Duration of Overall Response Rate | Baseline to measured progressive disease (up to approximately 12 months)
  Overall response was defined has having a response of Complete Response (CR) or Partial Response (PR). (See "Best Objective Tumor Response" Outcome Measure above for response category definitions.) Duration of Response is defined as the duration from the first overall response to the first Stable Disease (SD) or Disease Progression (PD), whichever happens first. If no SD or PD, subject is censored at the last tumor assessment (prior to other anti-cancer therapy if applicable).
Progression-free Survival (PFS) | Baseline to measured progressive disease (up to approximately 12 months)
  PFS was defined as the time from randomization to the date of disease progression or death, whichever occurred first, before or after treatment discontinuation. For participants still on study and those who remained alive and had not progressed after treatment discontinuation, PFS was censored on the date of the last tumor assessment.
Change From Baseline in Serum Hsp27 levels by End of Treatment | Baseline, End of Treatment (up to approximately 12 months)
  End of Treatment is last non-hemolyzed observation up to last dose + 30 days. Includes unscheduled and additional treatment visits. Hemolyzed samples were excluded.
Change From Baseline in Serum Clusterin Levels by End of Treatment | Baseline, End of Treatment (up to approximately 12 months)
  End of Treatment is last observation up to last dose + 30 days. Includes unscheduled and additional treatment visits.
Change From Baseline in Circulating Tumor Cell (CTC) Count by End of Treatment | Baseline, End of Treatment (up to approximately 12 months)
  End of Treatment is last observation up to last dose + 30 days. Includes unscheduled and additional treatment visits.
Serum OGX-427 Cmax and Trough Levels | Cycle 1 Day 1 through Cycle 6 Day 1, End of Treatment (up to approximately 12 months)
  only C1 to C6, Ctrough and Cmax - as well report EOT Ctrough

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Petrylak, MD, Principal Investigator — Columbia University
Locations (55):
- United States (14):
  - City of Hope National Medical Center, Duarte, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Radiological Associates of Sacramento, Sacramento, California
  - Yale University, New Haven, Connecticut
  - Karmanos Cancer Institute, Detroit, Michigan
  - Siteman Cancer Center, Washington University School of Medicine, St Louis, Missouri
  - Urology Cancer Center and GU Research Network, Omaha, Nebraska
  - Monter Cancer Center, Lake Success, New York
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, Albert Einstein College of Medicine, The Bronx, New York
  - Texas Oncology, P.A., Dallas, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
- Canada (7):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Cross Cancer Center, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - R. S. McLaughlin Durham Regional Cancer Center at Lakeridge Health, Oshawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUM-Hospital Notre Dame, Montreal, Quebec
- France (8):
  - Centre Hospitalier Régional et Universitaire - Hôpital, Bretonneau Tours, Centre-Val de Loire
  - Institute Jean Godinot, Reims, Champagne-Ardenne
  - Centre Hospitalier Universitaire de Rouen, Rouen, Haute-Normandie
  - Centre Paul Papin, Angers, Pays de la Loire Region
  - Medicale Centre René Gauducheau, Saint-Herblain, Pays de la Loire Region
  - Institut Paoli Calmettes, Marseille, Provence-Alpes-Côte d'Azur Region
  - Centre Antoine Lacassagne, Nice, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier Universitaire, Institut Gustave Roussy, Villejuif, Île-de-France Region
- Germany (9):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Klinikum Rechts der Isar der Technischen Universität, München, Bavaria
  - Johann-Wolfgang-Goethe-Universität Frankfurt, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Hanover, Niedeersachen
  - Universitätsklinikum des Saarlandes, Homburg, Saarland
  - Universitätsklinikum Dresden, Dresden, Saxony
  - Universitätsklinikum Magdeburg A.ö.R., Magdeburg, Saxony-Anhalt
  - Universitätsklinikum Jena, Jena, Thuringia
  - Universitätsklinikum Mainz, Mainz
- Italy (3):
  - Azienda Ospedaliero-Universitaria Policlinico di Modena, Modena
  - Fondazione IRCCS Policlinico San Matteo Pavia, Pavia
  - Unità Operativa di Oncologia Medica, Roma
- Poland (6):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Akademicki Szpital Kliniczny im. J. Mikulicza-Radeckiego we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - NZOZ Europejskie Centrum Zdrowia Otwock, Otwock, Masovian Voivodeship
  - Centrum Onkologii Instytut im. M. Sklodowskiej-Curie, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Zaklad Opieki Zdrowotnej MSWiA z Warminsko-Mazurskim Centrum Onkologii w Olsztynie, Olsztyn, Warminski-Mazurskie
- Spain (8):
  - Hospital Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Vall d´Hebrón, Barcelona
  - Institut Català D'Oncologia, Hospital Duran i Reynals, Madrid
  - Instituto Valenciano de Oncología-Fundación (IVO-FINCIVO), Valencia